CLINICAL TRIAL: NCT05887596
Title: The Effect of Patient Education on Pain Level and Fear of Pain in Orthopedians and Traumatology Patients
Brief Title: The Effect of Patient Education on Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Figen Calıskan, Associate Prof., Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/541
Record Dates: First submitted 2023-05-10; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Fear of Pain; Pain; Pain Management; Patient Education
Keywords: Fear of Pain; Pain; Pain Management; Patient Education
MeSH Terms: conditions — Pain; Agnosia | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The training given to the control group included preoperative preparation, operating theatre environment, breathing exercises, cough exercises, etc. to be performed after surgery. In both groups, temperature, pulse rate, blood pressure, oxygen saturation level, and pain level with a Visual/Visual Analogue Scale were measured on the morning of the operation day, before the operation, every 4 hours for 24 hours after the operation and on the day of discharge. Again, pain fear level was measured with the Fear of Pain Scale-III on the day of discharge in both groups.
- Intervention group (Experimental): The education given to the intervention group included preoperative preparation, operating room environment, breathing exercises, cough exercises, etc. to be performed after surgery, non-pharmacological methods related to pain management (cold application, positioning, distraction), and pharmacological methods related to pain management.
  Interventions: Other: Patient education

INTERVENTIONS:
Other: Patient education — The education given to the intervention group included preoperative preparation, operating room environment, breathing exercises, cough exercises, etc. to be performed after surgery, non-pharmacological methods related to pain management (cold application, positioning, distraction), and pharmacological methods related to pain management.
  Other Names: Patients receiving patient education on pain management
  Arms: Intervention group

SUMMARY:
Objective: The study was conducted to determine the effect of patient education on pain level and fear of pain in orthopedics and traumatology patients Methods: The study is a randomized controlled experimental research design. Data were collected between December 15, 2021, and March 15, 2022 using the Information Form, Fear of Pain Scale-III, and Visual/Visual Analogue Scale. A total of 52 patients, 26 in the intervention group and 26 in the control group were included in the study. The intervention group received patient education about the operation process and pain management the day before and the morning of the operation day. Number Cruncher Statistical System and Statistical Software (Kaysville, Utah, USA) were used to analyse the data Keywords: Fear of Pain, Pain, Pain Management, Patient Education

DETAILED DESCRIPTION:
Design The research is a randomized controlled experimental research design. Research hypotheses H1: The postoperative pain level of the patients in the intervention group is lower than that of the patients in the control group.

H2: The level of fear of postoperative pain of the patients in the intervention group is lower than that of the patients in the control group.

Research Variables Dependent Variables: Patients' pain level and fear of pain level Independent variable: Patient education Participants and setting The study group of the study consisted of 52 patients who underwent elective surgery in the orthopedics and traumatology clinic of the training and research hospital affiliated with the Ministry of Health in Istanbul between December 15, 2021, and March 15, 2022, and were open to communication and cooperation, had no cognitive and mental problems, and volunteered to participate in the study. The number of patients to be included in the study group; intervention and control were determined as a minimum of 25 patients (by calculating the margin of error of type 1 (α) = 0.05 and the power of the test (1-β) = 0.80, effect size 0.66 by power analysis of the patients constituting the universe). The study group consisted of a total of 52 patients, 26 in the intervention group and 26 in the control group, taking into account the possibility of data loss.

Intervention group: Patients receiving patient education on pain management Control group: Patients who did not receive training in pain management Patients who met the inclusion criteria were interviewed about the study. Patients who agreed to participate in the study were asked to choose an envelope containing an intervention or control letter. The patient with an intervention letter on the envelope was included in the intervention group and the patient with a control letter was included in the control group. Thus, bias in group selection was presented in the study.

Homogeneity between the groups was ensured by testing the gender, age, number of days of hospitalization, educational status, occupation, previous surgery, and regular use of pain medication. As a result of the analyses, it was found that there was no statistically significant difference between the gender, age, number of days of hospitalization, educational status, occupation, previous surgery, and regular use of pain medication in the intervention and control groups (p>0.05) (Table 1). According to the results, the intervention group (n: 26) and the control group (n: 26) showed homogenous distribution.

Data collection tools Data were collected using the Information Form, Fear of Pain Scale-III, and Visual/Visual Analogue Scale.

Information Form: The form, which was prepared by the researchers using the literature, includes 8 questions to determine the socio-demographic characteristics of the patients (gender, age, marital status, education level, occupation, number of days of hospitalization, previous surgery and regular medication use) (Büyükünal Şahin & Rızalar, 2018; Yang et al, 2019).

Fear of Pain Scale-III: The scale was developed by McNeil and Rainwater in 1998 to measure the fear of pain. The scale was adapted into Turkish by Ünver and Turan (2018). The scale consists of 30 items and 3 sub-dimensions "Fear of Severe Pain", "Fear of Mild Pain" and "Fear of Medical Pain" with 10 items in each sub-dimension. The response options of the scale prepared in 5-point likert type are; "5-extreme, 4-very much, 3-quite, 2-somewhat, 1-never". 1-never feeling fear, the 5-excessive feeling of fear. All items in the scale are positive and there are no reversed items. The lowest score that can be obtained from the scale is 30 and the highest score is 150. The minimum score for the sub-dimensions is 10 and the maximum score is 50. The higher the scores obtained from the scale, the higher the fear of pain. The total Cronbach alpha internal consistency coefficient of the scale is 0.93, 0.88 for the fear of severe pain sub-dimension, 0.85 for the fear of mild pain sub-dimension, and 0.93 for the fear of medical pain sub-dimension (Ünver & Turan, 2018).

Visual/Visual Analogue Scale: This scale is used to measure the level of pain. It is a one-dimensional scale. The scale is a 10 cm long ruler. It can be used horizontally or vertically. There are numbers from 0 to 10 on a scale of 0 (zero) "no pain" at one end and 10 (ten) "unbearable pain" at the other end. Pain level is measured by expressing the level of pain felt by the person with a numerical value from 0 to 10 (Eti Aslan & Yıldız, 2017).

Data collection The research was conducted between December 15, 2021, and March 15, 2022. Firstly, the patients to be included in the intervention and control groups were determined. Information Form, Fear of Pain Scale-III was applied to the patients in both groups, and pain levels of the patients were measured with the Visual/Visual Analogue Scale. Patients in the intervention group received patient education about the operation process and pain management the day before and on the morning of the operation day. Patients in the control group also received patient education about the operation process on the preoperative day and the morning of the operation day. The education given to the intervention group included preoperative preparation, operating room environment, breathing exercises, cough exercises, etc. to be performed after surgery, non-pharmacological methods related to pain management (cold application, positioning, distraction), and pharmacological methods related to pain management. The training given to the control group included preoperative preparation, operating theatre environment, breathing exercises, cough exercises, etc. to be performed after surgery. In both groups, temperature, pulse rate, blood pressure, oxygen saturation level, and pain level with a Visual/Visual Analogue Scale were measured on the morning of the operation day, before the operation, every 4 hours for 24 hours after the operation and on the day of discharge. Again, pain fear level was measured with the Fear of Pain Scale-III on the day of discharge in both groups. It took approximately 20-25 minutes to complete the data collection tools.

Data analyses Number Cruncher Statistical System (NCSS) 2007 Software (Kaysville, Utah, USA) was used for data analysis. Descriptive statistical methods (mean, standard deviation, median, frequency, percentage, minimum, maximum) were used. The conformity of quantitative data to normal distribution was tested by the Shapiro-Wilk test and graphical analyses. Independent groups t-test was used for comparisons of quantitative variables with normal distribution between two groups, and the Mann-Whitney U test was used for comparisons of quantitative variables without normal distribution between two groups. Pearson chi-square, Fisher's exact test, and Fisher-Freeman-Halton exact test were used in comparisons of qualitative data. Statistical significance was accepted as p<0.05 (Karagöz, 2014).

Ethical considerations Ethics committee approval was obtained from the Clinical Research Ethics Committee (Date: December 06, 2021 Number: 2021-23-14) of a training and research hospital (Bakirkoy Dr Sadi Konuk Training and Research Hospital). Institutional permission and permission to use the scale were obtained from the institution where the research would be conducted. Written informed consent was obtained from the patients included in the study.

ELIGIBILITY:
Inclusion Criteria:

* open to communication and cooperation,
* had no cognitive and mental problems,
* volunteered to participate in the study

Exclusion Criteria:

* closed to communication and cooperation,
* had cognitive and mental problems,
* not volunteered to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Pain Level | 3 months
  The primary point of the study was defined was assessed by a Visual/Visual Analogue Scale the effect of patient education on pain level in orthopedics and traumatology patients.

SECONDARY OUTCOMES:
Fear of Pain | 3 months
  The second point of the study was defined was assessed by the Fear of Pain Scale-III the effect of patient education on fear of pain in orthopedics and traumatology patients.

CONTACTS AND LOCATIONS:
Overall Officials: Figen Çalışkan, Assoc. prof, Principal Investigator — Trakya University, Turkey; Ayten Seller, Nurse, Principal Investigator — Bakırköy Dr. Sadi Konuk Training and Research Hospital, Turkey; Muhterem Gerçek, Nurse, Principal Investigator — Bakırköy Dr. Sadi Konuk Training and Research Hospital, Turkey
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caliskan F, Seller A, Gercek M. The Effect of Patient Education on Pain Level and Fear of Pain in Orthopedic Surgery: A Randomized Controlled Trial. J Perianesth Nurs. 2025 Jun;40(3):612-618. doi: 10.1016/j.jopan.2024.07.015. Epub 2024 Oct 24. PMID 39453348